CLINICAL TRIAL: NCT01868516
Title: Study Evaluating the Safety, Tolerability, and Efficacy of Dexmecamylamine (TC-5214) for Treatment of Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC-5214-23-CRD-003
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): One tablet of placebo to be administered orally twice a day.
  Interventions: Drug: Placebo
- 0.5 mg dexmecamylamine (TC-5214) (Experimental): One tablet of 0.5 mg dexmecamylamine to be administered orally twice a day.
  Interventions: Drug: dexmecamylamine
- 1 mg dexmecamylamine (TC-5214) (Experimental): One tablet of 1 mg dexmecamylamine to be administered orally twice a day.
  Interventions: Drug: dexmecamylamine
- 2 mg dexmecamylamine (TC-5214) (Experimental): One tablet of 2 mg dexmecamylamine to be administered orally twice a day.
  Interventions: Drug: dexmecamylamine

INTERVENTIONS:
Drug: dexmecamylamine
  Other Names: TC-5214
  Arms: 0.5 mg dexmecamylamine (TC-5214); 1 mg dexmecamylamine (TC-5214); 2 mg dexmecamylamine (TC-5214)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Overactive bladder (OAB) is a syndrome characterized by symptoms of a sudden need to urinate with or without incontinence (leaking). The purpose of this study is to test whether dexmecamylamine is safe and effective compared to placebo for the treatment of symptoms of OAB.

DETAILED DESCRIPTION:
The study included a three- or five-week screening period, followed by a 12-week treatment period during which patients received either one of three doses of dexmecamylamine or placebo twice daily, randomized in a ratio of 2:1:1:1 (placebo, low dose, mid dose, high dose), with a two-week follow-up period. A total of 768 subjects with overactive bladder were randomized into the double-blind treatment period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Verified medical history of overactive bladder for at least 6 months
* Capable of walking unassisted to use the bathroom
* Able to measure voided urine volume and complete the diary without assistance
* If the subject is currently being treated with an OAB medication, the subject is willing to discontinue OAB medications while participating in this study

Exclusion Criteria:

* Diagnosis of a neurological disease affecting bladder function
* Stress incontinence, insensate incontinence, overflow incontinence or incontinence due to urinary fistula
* History of incomplete bladder emptying, bladder outflow obstruction or post-void residual bladder volume > 150 mL
* Males with benign prostatic hyperplasia or with a prostate-specific antigen (PSA) of 4 ng/mL or more
* Other urinary tract pathology such as malignancy, ureteric reflux, bladder stone, uninvestigated hematuria, urethral stricture, or cystitis
* Prior treatment with intravesical or intraprostatic botulinum toxin in the last 2 years
* Myasthenia gravis
* Angle closure glaucoma
* Current implantation of interstim electrodes or vaginal surgical mesh
* Presence of a clinically significant medical condition at any time during the study
* Presence of clinically significant abnormalities in laboratory findings, physical exam findings or vital signs
* Participated in an investigational drug trial within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1635 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in micturition frequency per 24 hours | 12 weeks
  Micturition: Any voiding episode recorded by the patient as "urinated" either with or without incontinence.
Change from baseline in urinary urge incontinence (UUI) episodes per 24 hours | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the volume voided per micturition | 12 weeks
Change from baseline in nocturia per 24 hours | 12 weeks
  Nocturia: A micturition that wakes the subject from sleep between the time the subject went to bed and the time the subject woke up.
Clinical Global Impression of Improvement (CGI-I) | 12 weeks
Change from baseline in Patient Perception of Bladder Condition (PPBC) | 12 weeks
Change from baseline in the Urgency Questionnaire | 12 weeks
Change from baseline in disease specific quality of life (OABq) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (125):
- United States (125):
  - Simon-Williamson Clinic, P.C., Birmingham, Alabama
  - Physician's Resource Group, Dothan, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Mobile Ob-Gyn, P.C., Mobile, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Clinical Trials of Arizona, Inc., Glendale, Arizona
  - Beach Clinical Studies, Phoenix, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Atlantic Urology Medical Group, Long Beach, California
  - Adam D. Karnes, MD, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Northern California Research, Sacramento, California
  - San Diego Sexual Medicine, San Diego, California
  - Genesis Research, San Diego, California
  - Westlake Medical Research, Thousand Oaks, California
  - InFocus Clinical Research, Denver, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Meridien Reseach, Brooksville, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - 3H Clinical Research Corporation, Coral Springs, Florida
  - Palm Spring Research Institute, Hialeah, Florida
  - American Medical Research Institute, Kissimmee, Florida
  - Altus Research, Lake Worth, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Radiant Reseach, Inc., Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Perimeter North Medical Research, Inc., Roswell, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Radiant Research, Inc., Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - First Urology PSC, Jeffersonville, Indiana
  - Deaconess Clinic Gateway Health Center, Newburgh, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - GTC Research, Shawnee, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Bluegrass Clinical Research, Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Regional Urology, LLC, Shreveport, Louisiana
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Mid Atlantic Urology Associates, LLC, Greenbelt, Maryland
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Family Medicine Specialists, PC, Grand Rapids, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Westside Family Medical Center, PC, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saginaw Valley Medical Reseach Group, LLC, Saginaw, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Metro Urology, Woodbury, Minnesota
  - Mississippi Medical Research, LLC, Carriere, Mississippi
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Montana Health Research Institute, Inc., Billings, Montana
  - Five Valleys Urology, Missoula, Montana
  - Women's Clinical of Lincoln, P.C., Lincoln, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Lawrence OB-GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Delaware Valley Urology, LLC, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - SouthWest Clinical Research, Albuquerque, New Mexico
  - The Urological Institute of Northeastern New York, Albany, New York
  - Advanced Urology Centers of New York, Garden City, New York
  - Premier Medical Group of the Hudson Valley, PC, Kingston, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Radiant Research, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Physicians' Research, Inc., Zanesville, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Advanced Clinical Concepts, West Reading, Pennsylvania
  - Greater Providence Clinical Research, LLC, Warwick, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - Medical Research South, LLC, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - The Jackson Clinic, Jackson, Tennessee
  - Advanced Therapeutics, Inc., Johnson City, Tennessee
  - Tennesse Women's Care, Nashville, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - DiscoverResearch, Inc., Bryan, Texas
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Quality Research Inc., San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Reseach, Inc., San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - The Group for Women, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Inc., Norfolk, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Valley Women's Clinic, Renton, Washington
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington